CLINICAL TRIAL: NCT04970823
Title: The Effect of Somatosensory Interactive Games on the Pain, Fear and Negative Emotions of Children Receiving Intravenous Injection
Brief Title: The Effect of Interactive Games on Children Receiving Intravenous Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202012054RINC
Record Dates: First submitted 2021-06-30; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-01

CONDITIONS: Pain; Fear; Emotions
Keywords: school-age children; injection; pain; Somatosensory interactive games
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The somatosensory interactive game (Experimental): The somatosensory interactive game, an independent nursing intervention, promotes pain relief on the experimental group.
  Interventions: Device: The somatosensory interactive game for preschool children
- A VR (virtual reality) game (Experimental): A VR (virtual reality) game promotes pain relief on the experimental group.
  Interventions: Device: A VR (virtual reality) game for school-age children

INTERVENTIONS:
Device: The somatosensory interactive game for preschool children — The somatosensory interactive game, an independent nursing intervention, promotes pain relief for preschool children.
  Arms: The somatosensory interactive game
Device: A VR (virtual reality) game for school-age children — A VR (virtual reality) game environment promotes pain relief for school-age children.
  Arms: A VR (virtual reality) game

SUMMARY:
Pediatric intravenous injection is one of the most painful events that children may be exposed to during hospitalization or illness, and it is also the most routinely performed invasive procedure. The purpose of this study is to examine the effectiveness of somatosensory interactive games on intravenous pain relief for preschool children, and to establish a VR (virtual reality) game environment for school-age children. Using a randomized experimental study, the data came from the pediatric ward. The results will show whether there is a statistically significant difference between the experimental group and the control group.

DETAILED DESCRIPTION:
Pediatric intravenous injection is one of the most painful events that children may be exposed to during hospitalization or illness, and it is also the most routinely performed invasive procedure. Non-pharmaceutical techniques can be used to relieve pain associated with intravenous injections. Distraction is a non-pharmacological technique that can take child's attention away from pain. The somatosensory interactive game is an independent nursing intervention that promotes pain relief. The purpose of this study is to examine the effectiveness of somatosensory interactive games on intravenous pain relief for preschool children, and to establish a VR (virtual reality) game environment for school-age children. Using a randomized experimental study, the data came from the pediatric ward. At least qualified 132 preschool children are in this study and their caregivers signed a consent form to participate in the study. Children are divided into experimental group and control group, and each group has at least 66 children. In addition to 60 school-age children, 30 played VR games for about 3 minutes during intravenous injection, and 30 received regular intravenous injection. The preschool experimental group and the school-age experimental group each took the parents of 5 children (10 in total) to conduct semi-structured qualitative interviews to understand the differences in experience before and after the intervention. This study is expected to accept a total of 202 children and parents. Data collection tools include WBFPS (Wong-Baker Faces Scale) to measure children's pain and CFS (Children's Fear scale) to measure children's fear. CEMS continue assessment negative emotion two days. The results will show whether there is a statistically significant difference between the experimental group and the control group. Qualitative study used semi-structed interviews were conducted with selected and their parent.

ELIGIBILITY:
Inclusion criteria:

1. 2-7 years old, normal consciousness, preschool children who need intravenous injection.
2. 7-12 years old, normal consciousness, school-age children who need intravenous injection.
3. Parents of children need to be conscious and able to talk in Chinese.

Exclusion criteria:

1. 2-7 years old preschool children with developmental delay, epilepsy, heart disease, chemotherapy, visual and hearing impaired, obese, and have received more than 2 intravenous injections.
2. 7-12-year-old school-age children with developmental delay, epilepsy, heart disease, chemotherapy, visual and hearing impaired, obese, and have received more than 2 intravenous injections.
3. The child's parents cannot express and communicate effectively.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 202 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in children's pain from baseline to after intravenous injection | O1 (before intervention); O2 (immediately after intravenous injection); O3 (1 day after intravenous injection)
  Using Wong-Baker Faces Pain Rating Scale to measure pain. There are 6 faces in the Wong-Baker Pain Scale. The first face represents a pain score of 0, and indicates "no hurt". The second face represents a pain score of 2, and indicates "hurts a little bit." The third face represents a pain score of 4, and indicates "hurts a little more". The fourth face represents a pain score of 6, and indicates "hurts even more". The fifth face represents a pain score of 8, and indicates "hurts a whole lot"; the sixth face represents a pain score of 10, and indicates "hurts worst." Nurses, pre-school children by the assistance of caregivers, and school-age children were asked to evaluate the pain levels experienced by the children receiving intravenous injections.
Changes in children's fear from baseline to after intravenous injection | O1 (before intervention); O2 (immediately after intravenous injection); O3 (1 day after intravenous injection)
  Using Children's Fear scale to measure the fear level. Score the chosen face from 0 (the left-most face) to 4 (the last face). This face [point to the left-most face] shows no anxiety at all, this faces shows a little bit more [point to second face from left], a bit more [sweep finger along scale], right up to extreme anxiety [point to the last face on the right]. Nurses, pre-school children by the assistance of caregivers, and school-age children were asked to evaluate the fear levels experienced by the children receiving intravenous injections.
Changes in children's emotion from baseline to after intravenous injection | O1 (before intervention); O2 (immediately after intravenous injection); O3 (1 day after intravenous injection)
  Using Children's Emotional Management Scales to measure the emotion level. The scale includes five observed emotional behavior categories, facial expression, vocalization, activity, interaction, and level of cooperation. Each category is scored from 1-5 points, the lowest total score is 5 points, and the highest score is 25 points. The higher the score, the more negative emotional behavior. Nurses, pre-school children by the assistance of caregivers, and school-age children were asked to evaluate the emotion levels experienced by the children receiving intravenous injections.
semi-structed interviews | immediately after intravenous injection
  After intravenous injection, a semi-structured qualitative interview was conducted with selected and their parent to understand the differences in experience before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Mei Chen, OTHERS, Principal Investigator — NTUH Yunlin Branch
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan